CLINICAL TRIAL: NCT02763761
Title: A Phase 2, Randomized, Open-Label Study of Infliximab and Lower Exposure Corticosteroids vs Methylprednisolone and Higher Exposure Oral Corticosteroids for the Management of Immune-Related Severe or Persistent Diarrhea in Patients Treated With Yervoy (Ipilimumab) and/or Opdivo (Nivolumab)
Brief Title: An Investigational Study of Infliximab With Prednisone or Methylprednisolone Versus Prednisone Combination Treatment in Immune Related or Severe Diarrhea in Patients Treated With Yervoy and/or Opdivo
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-601
Record Dates: First submitted 2016-05-04; First posted 2016-05-05 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Renal Cell Carcinoma; Melanoma; Lung Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Melanoma; Lung Neoplasms | interventions — Infliximab; Prednisone; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Infliximab + Prednisone (Experimental): Infliximab intravenous solution (single dose) + low dose prednisone per oral for 18 days
  Interventions: Drug: Infliximab + Prednisone
- Methylprednisolone + Prednisone (Experimental): Methylprednisolone intravenous solution (single dose) + high dose prednisone per oral for 40 days
  Interventions: Drug: Methylprednisolone + Prednisone

INTERVENTIONS:
Drug: Infliximab + Prednisone — Prednisone dose will be decreased every 3 days for 18 days
  Arms: Infliximab + Prednisone
Drug: Methylprednisolone + Prednisone — Prednisone dose will be decreased every 4 days for 40 days
  Arms: Methylprednisolone + Prednisone

SUMMARY:
The purpose of this study is to compare the effects of Infliximab and oral prednisone versus methylprednisolone and oral prednisone in patients with melanoma, lung cancer, or renal cell carcinoma who have immune related Grade 3-4 diarrhea for up to 3 days or persistent Grade 2 diarrhea for more than 5 days after treatment with Yervoy and/or Opdivo

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Subjects must have melanoma or lung cancer or renal cell carcinoma and received ipilimumab or nivolumab as a single treatment or in combination
* Subject must have NCI common toxicity Grade 3-4 immune-related diarrhea for up to 3 days or persistent Grade 2 diarrhea for more than 5 days
* Subjects must be discontinued from ipilimumab or nivolumab as monotherapy or with the combination regimen

Exclusion Criteria:

* Subjects who received other anti Cytotoxic T-lymphocytic antigen (CTLA-4) (non-ipilimumab) or other anti-Programmed death-1 (PD-1) (non-nivolumab) treatment
* Subjects treated with systemic Corticosteroid (CST) within 1 week before randomization and subjects treated with infliximab within 7 weeks before randomization
* Subjects with known history of tuberculosis
* Subjects with immunosuppressive disease that require use of systemic steroids or immunosuppressive treatment
* Subjects allergic to infliximab, inactive components of infliximab, murine proteins and methylprednisolone

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08-16 (Actual); Primary Completion 2017-03-31 (Estimated); Study Completion 2017-03-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in management of immune related grade 3 and 4 diarrhea as measured by proportion of responders to less than or equal to grade 1 | Up to 78 hours
Improvement in management of persistent grade 2 diarrhea as measured by proportion of responders to less than or equal to grade 1 | Up to 78 hours

SECONDARY OUTCOMES:
Number of days to improvement to less than grade 1 diarrhea | Randomization up to 12 weeks
Quality of life as measured by European Quality of Life-5 Dimensions Questionnaire (EQ-5D) | Up to 12 weeks
Number of hospitalizations | Up to 12 weeks
Duration of hospitalizations | Up to 12 weeks
Number of patients with adverse events (AEs) | Up to 12 weeks
Number of patients with AEs related to steroid use | Up to 12 weeks
Number of patients with Gastrointestinal (GI) specific AEs | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (10):
- United States (10):
  - University of California Los Angeles, Los Angeles, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - University of Louisville, Louisville, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - Atlantic Health System, Morristown, New Jersey
  - Local Institution, Albuquerque, New Mexico
  - NYU Langone Medical Center, New York, New York
  - Huntsman Cancer Institute at The University of Utah, Salt Lake City, Utah

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx